CLINICAL TRIAL: NCT02176616
Title: Evaluation of Proper Radiofrequency Catheter Ablation Strategy for the Patients Who Were Changed to Paroxysmal Atrial Fibrillation From Persistent Atrial Fibrillation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4-2014-0279
Record Dates: First submitted 2014-06-23; First posted 2014-06-27 (Estimated); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- linear ablation (Active Comparator): The group of positive control is the operation to add in conventional liner ablation to conventional pulmonary vein isolation with in patients based on patients who were changed to paroxysmal atrial fibrillation from persistent atrial fibrillation
  Interventions: Procedure: linear ablation
- pulmonary vein isolation (Experimental): The group of negative is the operation to patients with only pulmonary vein isolation based on patients who were changed to paroxysmal atrial fibrillation from persistent atrial fibrillation
  Interventions: Procedure: pulmonary vein isolation

INTERVENTIONS:
Procedure: linear ablation — The group of positive control is the operation to add in conventional liner ablation to conventional pulmonary vein isolation with in patients based on patients who were changed to paroxysmal atrial fibrillation from persistent atrial fibrillation
  Arms: linear ablation
Procedure: pulmonary vein isolation — The group of negative is the operation to patients with only pulmonary vein isolation based on patients who were changed to paroxysmal atrial fibrillation from persistent atrial fibrillation
  Arms: pulmonary vein isolation

SUMMARY:
1. Purpose of the study

1) To compare clinical outcome, procedure time, complication rate of patients who were changed to paroxysmal atrial fibrillation from persistent atrial fibrillation between ablation with conventional pulmonary vein isolation and ablation with conventional pulmonary vein isolation with conventional linear ablation.

2. Scientific evidence of the study

1. In atrial fibrillation patients, the maintenance of normal sinus rhythm showed significant reduction of mortality.
2. drug therapy with anti-arrhythmic drug showed many complications and side effect, thus non-drug therapy such as catheter ablation is developed.
3. catheter ablation has been performed for 10years world-wide, and showed superior treatment outcome compared with drug therapy.
4. However, there are no consensus for proper ablation strategy in patients who were changed to paroxysmal atrial fibrillation from persistent atrial fibrillation .
5. additional ablation make extent of myocardial injury and paradoxically increase recurrence rate, thus still controversial.
6. Therefore, we will compare conventional pulmonary vein isolation with additional conventional linear ablation.

3. Methods

1. Treatment of All patients with atrial fibrillation is performed according to the standard treatment guideline of atrial fibrillation.
2. there is no additional blood sampling, imaging study, or any other invasive procedure according to the inclusion of the study.

4. study contents

1) to evaluate superior ablation strategy in patients who were changed to paroxysmal atrial fibrillation from persistent atrial fibrillation

* compare conventional pulmonary vein isolation with additional liner ablation, both strategies are conventional ablation strategies being performed world-wide.

ELIGIBILITY:
Inclusion Criteria:

1) patients who undergoing catheter ablation of atrial fibrillation due to symptomatic, drug refractory atrial fibrillation

Exclusion Criteria:

1. patients who do not agree with study inclusion
2. permanent AF refractory to electrical cardioversion
3. AF with valvular disease ≥ grade 2
4. Patients with left atrial diameter greater than 60mm
5. patients with age less than 19

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2014-06; Primary Completion 2024-02 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
number of Clinical recurrence of atrial fibrillation (AF) after catheter ablation | 1 year
  lifelong, checked per every outpatient clinic visit

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Pak HN, Park J, Park JW, Yang SY, Yu HT, Kim TH, Uhm JS, Choi JI, Joung B, Lee MH, Kim YH, Shim J. Electrical Posterior Box Isolation in Persistent Atrial Fibrillation Changed to Paroxysmal Atrial Fibrillation: A Multicenter, Prospective, Randomized Study. Circ Arrhythm Electrophysiol. 2020 Sep;13(9):e008531. doi: 10.1161/CIRCEP.120.008531. Epub 2020 Jul 28. PMID 32755396
- [Derived] Yu HT, Shim J, Park J, Kim IS, Kim TH, Uhm JS, Joung B, Lee MH, Kim YH, Pak HN. Pulmonary Vein Isolation Alone Versus Additional Linear Ablation in Patients With Persistent Atrial Fibrillation Converted to Paroxysmal Type With Antiarrhythmic Drug Therapy: A Multicenter, Prospective, Randomized Study. Circ Arrhythm Electrophysiol. 2017 Jun;10(6):e004915. doi: 10.1161/CIRCEP.116.004915. PMID 28611206